CLINICAL TRIAL: NCT05919056
Title: Cardiovascular Risk Assessment and dynamIc Monitoring-based Prevention Trial for prImary Care quALity evaLuation in Yinzhou
Brief Title: Cardiovascular Risk Assessment and Dynamic Monitoring-based Prevention Trial
Acronym: CRITICALLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Yinzhou District Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Pei Gao, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00001052-21060
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases
Keywords: primary prevention; cluster randomized trial; cardiovascular risk assessment
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The interventions include cardiovascular risk assessment, dynamic risk monitoring, and regular general practitioner (GP) visits. The frequency of risk assessment, risk monitoring, and automatic mobile texting will be once per month, while regular GP visits will be once per three months.
  Interventions: Other: Frequent and automatic cardiovascular risk assessment; Other: Dynamic risk monitoring; Other: Regular GP visits
- Control arm (No Intervention): Current regular management (usual care) will be kept in the control arm. The management objectives are for patients with hypertension or diabetes mellitus. The frequency of follow-up is at least once per three months.

INTERVENTIONS:
Other: Frequent and automatic cardiovascular risk assessment — The 10-year cardiovascular risk scores using the 2019 World Health Organization (WHO) laboratory-based risk charts will be automatically calculated using the latest health information on an EHR-based system per month.
  Arms: Intervention arm
Other: Dynamic risk monitoring — High-risk individuals will be reassessed by the Dynamic Risk-based Early wArning and Monitoring (DREAM) system to obtain the short-term risk. The DREAM system will send a text message about advice to the high-risk individual every month. The text message includes information on the health status (e.g., current cardiovascular risk, level of blood pressure and lipid) and real-time warning messages (e.g., high short-term risk).
  Arms: Intervention arm
Other: Regular GP visits — The general practitioners will communicate with the participants based on the information automatically generated from the DREAM system every three months: each participant's cardiovascular risk score, health status (e.g., diabetes mellitus and/or hypertension), and Chinese guidelines-based recommendations (e.g., "for the management of dyslipidemia, to provide clear treatment targets for high-risk participants").
  Arms: Intervention arm

SUMMARY:
The CRITICALLY study is a cluster randomized trial that will evaluate the effectiveness of a risk-based dynamic monitoring strategy for the primary prevention of cardiovascular high-risk Chinese adults.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the effectiveness of a risk-based management strategy on cardiovascular risk scores (calculated by the 2019 WHO cardiovascular risk charts) in 24 months (Phase I) and the incidence of major adverse cardiovascular events in 60 months (Phase II). Totally 216 clinics in Yinzhou District, China will be randomized to the intervention or the control arms with usual care. The interventions supported by the web-based decision support system include (1) cardiovascular risk assessment, (2) dynamic risk monitoring, and (3) regular visits by the general practitioner every three months. Only usual care will be provided in the control arm. The primary outcome is the change in cardiovascular risk scores for Phase I and the incidence of the composite endpoint of coronary heart disease, stroke, heart failure and all-cause mortality for Phase II. If the comprehensive strategy is proven effective, it could provide evidence for the primary prevention of cardiovascular diseases using digital health technology.

ELIGIBILITY:
Inclusion Criteria:

* Residents in the Yinzhou District have a unique health ID;
* Aged 40 to 79 years at the baseline enrollment;
* With high risk of cardiovascular disease evaluated by the 2019 WHO laboratory-based risk models (10-year risk≥10%);

Exclusion Criteria:

* Have a history of coronary heart disease, stroke or heart failure;
* Patients with a diagnosis of cancer;
* Refused to provide written informed consent

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22032 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome of Phase I: Change in cardiovascular risk score | 24 months after baseline
  The change in cardiovascular risk scores calculated by 2019 WHO laboratory-based risk charts
Primary Outcome of Phase II: Major adverse cardiovascular events (MACE) | 60 months after baseline
  Incidence of coronary heart disease, stroke, heart failure and all-cause mortality

SECONDARY OUTCOMES:
Secondary Outcome of Phase I: Change in systolic blood pressure | 24 months after baseline
  the change in systolic blood pressure from baseline
Secondary Outcome of Phase I: Change in total cholesterol | 24 months after baseline
  the change in total cholesterol from baseline
Secondary Outcome of Phase I: Change in low-density lipoprotein cholesterol | 24 months after baseline
  the change in low-density lipoprotein cholesterol from baseline
Secondary Outcome of Phase II: Change in health-related quality of life | 60 months after baseline
  Measured using the EuroQol-5 Dimensions-5L(EQ-5D)

OTHER OUTCOMES:
Other Pre-specified Outcome of Phase II: Incremental cost-effectiveness ratio (ICER) | 60 months after baseline
  the incremental cost-effectiveness ratio (ICER) of the management provided by the interventions compared to the usual care

CONTACTS AND LOCATIONS:
Overall Officials: Xun TANG, PhD, MHS, Principal Investigator; Pei GAO, PhD, Principal Investigator
Locations (1):
- Yinzhou District Center for Disease Control and Prevention, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
According to the Administrative Regulations on Human Genetic Resources issued by the State Council of the People's Republic of China in 2019, we are waiting for the approval of IPD sharing.

REFERENCES:
- [Background] Lin H, Tang X, Shen P, Zhang D, Wu J, Zhang J, Lu P, Si Y, Gao P. Using big data to improve cardiovascular care and outcomes in China: a protocol for the CHinese Electronic health Records Research in Yinzhou (CHERRY) Study. BMJ Open. 2018 Feb 12;8(2):e019698. doi: 10.1136/bmjopen-2017-019698. PMID 29440217
- [Background] Liu XF, Li QQ, Chen WY, et al. A dynamic risk-based early warning monitoring system for population-based management of cardiovascular disease. Fundamental Research. 2021:534-542.
- [Background] Liu X, Shen P, Zhang D, Sun Y, Chen Y, Liang J, Wu J, Zhang J, Lu P, Lin H, Tang X, Gao P. Evaluation of Atherosclerotic Cardiovascular Risk Prediction Models in China: Results From the CHERRY Study. JACC Asia. 2022 Jan 4;2(1):33-43. doi: 10.1016/j.jacasi.2021.10.007. eCollection 2022 Feb. PMID 36340248